CLINICAL TRIAL: NCT06294379
Title: Shared Decision Making in Melanoma Patients Receiving Adjuvant Therapy: Development of a Decision Aid Tool
Brief Title: Shared Decision Making in Melanoma Patients Receiving Adjuvant Therapy
Status: Recruiting | Type: Observational
Sponsor: Odense University Hospital (Other)
Collaborators: University of Copenhagen (Other); Aarhus University Hospital (Other); Aalborg University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: OUH_SDM
Record Dates: First submitted 2023-12-19; First posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-02

CONDITIONS: Malignant Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to develop test and evaluate a Patient Decision Aid called "The Decision Helper" among melanoma patients eligible for adjuvant treatment.

* Is the Decision Helper an acceptable tool for patients and clinicians and is it feasible in clinical practice?
* Are there any differences in the levels of decisional regret in the patients who have not used the Decision Helper (pre-implementation) compared to the ones who have (post-implementation?

DETAILED DESCRIPTION:
Malignant Melanoma Worldwide, the incidence of melanoma of the skin continues to increase. Cutaneous melanoma is the most lethal skin cancer worldwide. In alignment with the global trend, the number of Danes who are diagnosed with malignant melanoma has also increased significantly during the last 50 years. In Denmark, approximately 400 persons are diagnosed with metastatic disease each year. Although more people are diagnosed with melanoma, there has only been a minor increase in the number of people who die from the disease. This is primarily due to improved treatment modalities. The development of immunotherapy and targeted therapy have been the most important breakthroughs in melanoma treatment. In the last decade, immune checkpoint inhibitors (CPIs) have improved survival significantly for patients with metastatic melanoma. However, the immune-related adverse events (irAEs) that patients may experience can be severe and potentially life-threatening.

Adjuvant therapy When it comes to the treatment of malignant melanoma, it is not only in the metastatic setting that treatment options have improved disease control. The scene has also changed when it comes to adjuvant treatment where CPIs also play an increasingly important role. Until recently, the standard of care after completely resected stage III melanoma was active surveillance. In stage III melanoma the cancer has spread from the skin cells to the lymph nodes, which means that these patients are considered to have a high risk of recurrence; a part of them will at some point experience a relapse with metastatic disease. Consequently, several drugs to prevent recurrence after surgery have been tested in melanoma over the years, but until recently none had proven effective. The first drug to change this was the CPI, Ipilimumab. In 951 patients with resected melanoma at high risk of recurrence stage (IIIa, IIIb, or IIIc disease), the effectiveness of Ipilimumab as adjuvant therapy was tested. The recurrence-free survival was significantly improved in favor of the patients who had received Ipilimumab compared with placebo. 5-year rate of recurrence-free survival was 41% in the ipilimumab group, as compared with 30% in the placebo group. However, more than half of the patients experienced severe irAEs. Ipilimumab was never approved as a standard adjuvant treatment in Denmark due to the high risk of severe irAEs. However, in December 2018 two other CPIs, Nivolumab and Pembrolizumab, were approved as adjuvant treatment (for stage IIIa, IIIb, or IIIc resected disease). Nivolumab has proved to increase recurrence-free survival when compared to ipilimumab. 4-year recurrence-free survival was 52% in the Nivolumab group and 41% in the ipilimumab group. In addition, only around 14% of the patients who receive monotherapy with Nivolumab experience a grade 3 or 4 adverse events (AE). Similar results were found in another study investigating the CPI, anti-PD1 antibody, Pembrolizumab. The overall risk of recurrence was reduced by approximately 40% across stages as a result of adjuvant therapy with Pembrolizumab after 3 years [12]. Despite the gain in recurrence-free survival, there I not always a best/right decision regarding adjuvant treatment. In the following the pros and cons for starting adjuvant treatment will be described in more detail, illustrating the inherent dilemma between clinical benefit and irAEs.

The challenges of adjuvant therapy - to treat or not to treat There is prognostic heterogeneity within the group of stage III melanoma patients. The risk of experiencing a relapse varies depending on whether a patient is diagnosed with stage IIIA disease or stage IIIC disease (AJCC 7th Edition). Thus, some patients have a low risk of recurrence, (stage IIIA), while others are at greater risk (stage IIIC) following complete resection.

Patients with stage IIIC also have more to gain from a prognostic perspective than patients with stage IIIA disease if they receive adjuvant treatment. Even though all patients with stage III disease are eligible for adjuvant therapy, the decision to initiate treatment is not unproblematic. Furthermore, the number of melanoma patients who are candidates for adjuvant treatment is likely to increase in the future. Randomized controlled trials are currently investigating if patients with stage IIB/C melanoma can also benefit from adjuvant therapy. The argument is that these patients have a prognosis similar to patients with stage IIIB melanoma.

In addition to the fact that some patients are considered to be at low risk of relapse, there is also the question of toxicity. Almost 80% of the patients who receive adjuvant immunotherapy experience some kind of irAE, and approximately 14% of the patients experience severe irAEs that in some cases can be fatal.

Moreover, severe toxicities can impact patients´ quality of life. O´Reilly et al conclude in a paper published in 2019 that melanoma patients who had received immunotherapy have potentially experienced significant irAEs during treatment resulting in chronic conditions and exposure to significant doses of steroids. Accordingly, they had significantly lower health-related quality of life scores about physical, social, and physical role functioning and general health compared with healthy controls. Moreover, if/when patients relapse with metastatic disease, they are often offered treatment with the same drug as they would have received in the adjuvant setting, which may support the argument that some of the patients are better off waiting. On the other hand, patients of course prefer not to have a relapse. Thus, there is not always an obvious best treatment and the decision to treat or not to treat can be challenging. It is currently not well understood how patients eligible for adjuvant immunotherapy make their decision to accept or not accept treatment, and careful consideration and discussion about the potential risks and benefits must be carried out with each patient. In addition to disease recurrence, physicians must keep several factors in mind such as patient age, comorbidity, and personal preferences.

Patient involvement As it is impossible to predict which patients will benefit from the treatment, international guidelines developed for other patient populations suggest that adjuvant systemic treatment, particularly in cases where there is little to gain (for example patients with stage IIIA disease), should be discussed with the patient. This recommendation to include the patients when it comes to decisions about treatment and care is in line with the general trend within the health care system. The Danish National Survey of Patient Experiences (LUP) stresses that the dimension "patient involvement" is the most poorly rated area of all dimensions rated by the patients in the survey. Moreover, the Region of Southern Denmark decided in 2019 that Shared Decision Making (SDM) should be deployed in all hospitals in the region. Thus both politicians as well as patient organizations have an increased focus on involving the patients more engagement.

Shared Decision Making - a possible game changer According to the Danish Melanoma Group, approximately 100 patients are eligible for adjuvant treatment annually at the Department of Oncology, Odense University Hospital. Patients and physicians face the difficulties described above, when having to decide which melanoma patients are to receive adjuvant therapy. Sometimes the choice may seem obvious because the patients may have a relatively high risk of recurrence. In other situations where the patients have a low risk of recurrence or comorbidities which may make treatment with immunotherapy risky, it is more complex. In such cases, SDM could be useful to support this preference-sensitive decision. SDM is defined as "an approach where clinicians and patients share the best available evidence when faced with the task of making decisions, and where patients are supported to consider options, to achieve informed preferences and in making treatment decisions that align with these preferences". A Danish lung cancer study from 2019 showed that patients who had been engaged in SDM had lower decisional conflict and regret. Furthermore, they felt more confident about the decision and the process facilitated that patients´ values played a more central role in decision-making. One way to increase the level of patient-perceived involvement and make the consultations in the outpatient clinic more uniform may be to use a patient decision aid (PtDA) to support shared decision-making. If the patients experience that they are part of the decision process, it may also result in a lower level of decisional regret as described above.

Patient Decision Aids In other countries such as the United States decision-support tools have been developed, containing information on what the patients need to know about stage III melanoma. The patients can find information about the disease, substages, adjuvant therapy vs active surveillance, side effects, and outcomes. With this information in mind, the patients may be able to weigh the options with their treating oncologist to come to the right decision. Only a few decision aids have been developed and tested scientifically in a Danish context. As mentioned, adjuvant therapy as standard treatment is a relatively new treatment option for patients with melanoma, and no recipe guides/describes how to reach the right shared decision for the individual patient. However, a study carried out in oncology care and pulmonary medicine demonstrates how the use of a patient decision aid (PtDA) enhanced SDM in two different settings and helped increase focus on patient preferences [25]. This study used a generic patient decision aid template, called "Decision Helper" developed by the Center for Shared Decision Making in the Region of Southern Denmark (CFFB). Therefore, the center now offers a platform for decision-aid templates that adhere to the certification and quality criteria set by the International Patient Decision Aid Standards (IPDAS). Utilizing log-in, healthcare providers have access to the platform and the template for building patient decision aids (BESLUTNINGSHJÆLPER™) and will be able to build and develop PtDAs tailored to their specific needs. The template is developed based on the IPDAS criteria.

Study 1 - Development of the Patient Decision Aid

Methods: As both patients and clinicians are the end-users of the PtDA, both groups will participate in an iterative process to ensure that patient needs are prioritized and that the PtDA is relevant, accurate, and easy to use. Thus, instead of just seeing the patients as a source of data, they will play an active role in the design phase of the PtDA. A qualitative approach will be applied using semi-structured interviews, as recommended in IPDAS guidelines, where melanoma patients and clinicians will identify the type and amount of information needed for creating relevant and appropriate PtDA. As a supplement to this, another qualitative method (observational) will be used as a researcher (the project manager) will observe the patient-clinician communication (before the introduction of the PtDA) in a natural situation to collect data on the communication between the patient and clinician, how the talk is organized and the level of patient involvement.

Phase 1: Preparation of the Patient Decision Aid

* Observation by researcher in the outpatient clinic - 5 consultations
* An expert group consisting of physicians and nurses will look at PROs and CONs for receiving treatment/not receiving treatment
* Interviews with melanoma patients, who have already decided whether to receive treatment or not, about their views and preferences and what they see as advantages and disadvantages. An interview guide will be prepared to ensure uniformity and all aspects are covered. Three patients who have accepted treatment and three patients who have declined will be included.

Phase 2: Design of the Patient Decision Aid

The PtDA will be prepared following the views and preferences of patients and clinicians with the following content:

* Introduction: It must be clear to the patients that a PtDA is used in the consultation for the patient and the clinician to make a decision together
* The choices must be clear to the patient (observation or treatment)
* Focus on patient preferences - what matters to the patient
* Description of the different choices using 4 cards describing:

  * PROs and CONs/risks and benefits
  * Patient stories (patients who have made the choice already, see phase 1)
  * Statistics (risk of relapse)
  * Timeline (Description of the trajectory for both choices (treatment or observation).

Data entered into IT platform 1. Draft prepared Information/data from phase 2 is entered into the IT platform BESLUTNINGSHJÆLPER and the first draft is ready. The Center of Shared Decision-Making will provide support and feedback.

User test - 2. draft prepared A user test is carried out, including individual interviews with 3-4 patients and 3-4 clinicians. For the patients, a semi-structured interview guide will be used that is based on the items from the Preparation for Decision-Making Scale. Similarly, a guide will be prepared for clinicians. Based on the findings from the interviews and usability testing, the decision helper will be refined, and changes will be entered into the IT platform.

Trial period - 3. draft prepared The final version is printed and a trial period of approximately 12 weeks will take place. If no further adjustments are required, the PtDA is ready for implementation.

Study 2 - Evaluation of the PtDA Hypothesis: The implementation of the PtDA will result in an increased level of patient involvement among melanoma patients eligible for adjuvant immunotherapy. In addition, the patients will experience less decisional regret. Moreover, the consultations in the outpatient clinic will become more uniform and consistent.

Aims: To investigate 1)the level of patient involvement and 2)decisional regret among melanoma patients receiving adjuvant therapy before and after implementation of the PtDA. In addition, 3) to examine if the consultations become more uniform and consistent.

Methods: Since the aim was to examine the level of patient involvement, decisional regret, and the uniformity and consistency of consultations before and after the implementation of the PtDA, it has been decided to use a pre-post study design. Although this design does not take other factors that may change during the study into account, it may be able to suggest if the outcome is impacted by the intervention. A mixed method approach will be used to evaluate the effect of the PtDA, using both quantitative data and the Decision Regret Scale) and qualitative data (individual interviews and focus group interviews.) A convergent design is selected, in which survey data and interview data are collected in parallel over the same period. This will be described in more detail for each of the three aims in the following.

- Level of patient involvement Qualitative data: The level of patient involvement will be examined using a qualitative approach, by conducting interviews with eligible patients before and after implementation. Due to the exploratory nature of the study, the sample size cannot be determined in advance, but the aim is to include 10-15 patients for both pre and post-interviews depending on when data saturation has been reached. A purposive sample of patients will be selected to ensure maximal variation in gender, age, and treatment choice. A semi-structured interview guide will be designed to make the interaction as smooth as possible and the interviews will carried out by the same interviewer to ensure uniformity. Members of the project group will participate in the coding and analysis of the interviews. Braun and Clarke six step theory will be used for analysis.

Quantitative data:

Qualitative data: Focus group interviews will be carried out with clinicians who take part in outpatient consultations before and after implementation to elucidate if the consultations have become more uniform and consistent after the inclusion of the PtDA. Due to the limited number of physicians and nurses caring for/treating the patient population, it will only be possible to carry out two focus group interviews before and after. The interviews will consist of approximately 5-6 clinicians each. As with the individual interviews, an interview guide will be prepared and the interviews conducted in a semi-structured manner. The same content analysis approach will be applied to the group interview as described above.

Quantitative data: The plan is to measure the time spent on the individual consultation to elucidate if the time consumption differs between the two groups i.e. if the length of the consultations has been more uniform after implementation.

- Decision regret Quantitative data: Patients who have not been exposed to SDM (pre-implementation) and patients who have been exposed (post-implementation) will be asked to complete the Decision Regret Scale (DRS). The DRS is a questionnaire that measures distress and remorse after a healthcare decision. The scale consists of 5 questions. The scores are converted into a 0-100 scale following the user manual. A score of 0 means no regret; a score of 100 means high regret.

Statistics:

Primary outcome: DRS (0-100 scale, 20 steps), mean before/after compared by linear regression with bootstrapped standard errors (To take into account non-normality of scores). Secondary analysis: Tested with Wilcoxon rank-sum test Secondary outcomes: DRS above cutoffs for mild (5-25), respectively, moderate/strong regrets (≥ 30): Compared by logistic regression.

Supplementary analysis: In supplementary analyses above regressions will be adjusted for patient characteristics, which might have changed between the before and after periods.

Sample size calculations:

Collaborators The study is supported by the head of department at the Department of Oncology at Odense University Hospital. Two patient representatives and the team (physicians and nurses) that is responsible for the treatment will play a vital part in developing the PtDA to ensure that all aspects are covered. Furthermore, the study will be carried out in collaboration with "The Center for Shared Decision-Making". Finally, a cross-sectional survey, including various questionnaires, was sent out to 427 melanoma patients across Denmark in March this year. The Decision Regret Scale (DRS) is one of the questionnaires in the survey and accordingly, it will be elucidated if the patients who have received adjuvant treatment in 2019 and 2020 have had any decisional regret. The results will be helpful as historical background data for our project.

Perspectives The studies will be based at the Department of Oncology, OUH, but the project is highly relevant for all melanoma patients in Denmark. It is expected to change how outpatient consultations take place, enabling the patients to participate in important decision-making regarding their treatment and care. It is currently not well understood how patients eligible for adjuvant immunotherapy make their decision to accept or not accept treatment. It is expected that the PtDA for melanoma patients receiving immunotherapy in the adjuvant setting can be used nationwide and serve as an example for other researchers/clinicians who wish to design a similar tool for other patient populations receiving immunotherapy. Moreover, because the researchers also aim to evaluate the tool by comparing the level of patient involvement before and after implementation of the "Decision Helper", it will be elucidated if the designed tool makes a difference.

ELIGIBILITY:
Inclusion Criteria:

* Danish speaking
* Diagnosed with stage 3 malignant melanoma
* Eligible for adjuvant immunotherapy

Exclusion Criteria:

* Metastatic disease
* Mental impairment

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with malignant melanoma who at about to receive adjuvant therapy with immunotherapy or targeted therapy
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Development of a Patient Decision Aid "The Decision Helper" for melanoma patients receiving adjuvant theory | 1 year
  To develop a Patient Decision Aid for melanoma patients receiving adjuvant theory
Evaluation of the "The Decision Helper" | 1 year
  To evaluate "The Decision Helper among patients and healthcare professionals"

CONTACTS AND LOCATIONS:
Locations (1):
- Odense University Hospital, Odense C, Denmark